CLINICAL TRIAL: NCT06650254
Title: Investigation of the Effect of Structured Breastfeeding Support Based on Kolcaba's Comfort Theory on Breastfeeding Comfort of Mothers
Brief Title: Investigating the Effect of Breastfeeding Support on Mothers Breastfeeding Comfort
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge Kaya (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Ozge Kaya, Lecturer, İstanbul Yeni Yüzyıl Üniversitesi
Organization: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Özge KAYA
Record Dates: First submitted 2024-09-06; First posted 2024-10-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breastfeeding Support
Keywords: Kolcaba's Comfort Theory; Breastfeeding; Breastfeeding Support; Breastfeeding Comfort
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single blind (researchers are not blinded) randomization is recorded as the mothers will be supported by the researchers face to face and via the Web application. The statistician is also blinded for data analysis purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The mothers in the control group will be followed in line with the hospital's routine health monitoring and information.
- Breastfeeding Support Program Structured According to Kolcaba's Comfort Theory (Experimental): Mothers who are on postpartum day 0 will be included in the "Breastfeeding Support Program Structured According to Kolcaba's Comfort Theory" in addition to the routine follow-up and training they can receive from the hospital.
  Interventions: Other: Breastfeeding Support Program Structured According to Kolcaba's Comfort Theory

INTERVENTIONS:
Other: Breastfeeding Support Program Structured According to Kolcaba's Comfort Theory — Stage 1: The "Postpartum Breastfeeding Comfort Scale" will be applied to mothers before they are admitted to the support program. On the 0th day postpartum, the researcher will go to the mother, baby and father and provide "mother-baby skin-to-skin contact and breastfeeding support (Module 1)".
  Stage 2: The videos aimed at increasing breastfeeding comfort, which were shot for Modules 2, 3, 4 and 5 and transferred to the website, will be watched by mothers and fathers/relatives after discharge. At the same time, online counseling will be provided through the website and support will be provided for applications that will increase breastfeeding comfort.
  Stage 3: Mothers who have participated in at least 70% of the breastfeeding support structured according to Kolcaba's Comfort Theory will be called after 6-8 weeks and the "Postpartum Breastfeeding Comfort Scale" will be applied again and their final tests will be performed.
  Arms: Breastfeeding Support Program Structured According to Kolcaba's Comfort Theory

SUMMARY:
The World Health Organization and the United Nations Children's Fund report that exclusive breastfeeding for six months and continuing breastfeeding for two years or longer with appropriate complementary foods is one of the most powerful practices to increase the survival and well-being of the child. Some difficulties experienced during the breastfeeding process negatively affect the continuation of breastfeeding and prevent the baby from receiving breast milk. It has been determined in the studies in the literature that various interventions have been made and recommendations have been made to increase breastfeeding rates. However, it has been seen that there is a need for studies that address the needs of mothers regarding breastfeeding problems in a holistic manner and provide support in line with their needs. In order to increase breastfeeding success and ensure the continuity of effective breastfeeding, it is obvious that a holistic assessment of mothers; breastfeeding problems is needed, physical, psychospiritual, sociocultural and environmental factors that may cause deterioration in comfort are determined and comfort-focused nursing support is provided. In this context, the aim of the study is to determine the effect of the breastfeeding support structured according to Kolcaba's comfort theory given to mothers in the postpartum period on the breastfeeding comfort of mothers, and the second aim is to develop the "Postpartum Breastfeeding Comfort Scale" and test its validity and reliability.

Hypotheses of the study:

H0: The breastfeeding support structured according to Kolcaba's comfort theory given to mothers in the postpartum period is not an effective method in increasing the breastfeeding comfort of mothers.

H1: The breastfeeding support structured according to Kolcaba's comfort theory given to mothers in the postpartum period increases the breastfeeding comfort of mothers.

H2: "Postpartum Breastfeeding Comfort Scale" is a valid and reliable tool for measuring mothers' breastfeeding comfort.

DETAILED DESCRIPTION:
Breastfeeding is a safe, clean, healthy and easily accessible form of nutrition under all circumstances. Breastfeeding supports the immune system of babies, reduces mortality and morbidity rates, and reduces the risk of chronic diseases such as obesity and diabetes in later life. Breastfeeding also has a positive effect on maternal health, reducing the risk of breast and ovarian cancer, type 2 diabetes and hypertension. Thanks to breastfeeding, bonding behavior develops between the newborn and the mother, which makes the mother feel more successful. The World Health Organization has reported that the rate of exclusive breastfeeding for the first 6 months should be at least 50% as the 2025 target, and this rate should be at least 70% by 2030. Despite all these benefits of breastfeeding and the recommendations of the World Health Organization, 48% of babies aged 0-5 months worldwide are exclusively breastfed. While South Asia is the region where babies are most commonly exclusively breastfed with 60% of their babies, only 26% of babies aged 0-5 months are exclusively breastfed in North America. In our country, according to the 2018 Turkey Demographic and Health Survey, only 41% of babies under six months are breastfed, and the intake of only breast milk drops to 59% in the first month, 45% in the second and third months, and 14% in the fourth and fifth months.

Some difficulties experienced during the breastfeeding process negatively affect the continuation of breastfeeding and prevent the baby from receiving breast milk. In a mixed method study conducted to identify breastfeeding problems experienced in the early period, they reported that nearly 40% of mothers had breastfeeding problems in the early period and that the problems were due to lack of support from the mother-baby and health professionals. It was observed that the baby not being able to latch on to the breast (40%) and the mothers nipples being sore, injured, and cracked (38%) were the prominent problems. Conducted an observational study involving 552 mothers to investigate the breastfeeding difficulties experienced by mothers in the first months after birth and their relationship with early cessation of breastfeeding. They found that approximately 70.3% of mothers experienced problems such as breastfeeding difficulties, reporting cracked nipples, insufficient perception of milk quantity, pain and fatigue. They reported that the difficulties mostly occurred in the first month and emphasized that continuous, personalized professional breastfeeding support is very important based on the study results.

In a systematic review conducted to examine the effects of interventions on the nipple and breastfeeding in cases of flat and/or sunken nipples, which frequently cause mothers to stop breastfeeding early, it was reported that the Hoffman exercise, the reverse syringe method and nipple exercise were highly effective in increasing breastfeeding success, and that the rates of exclusive breastfeeding in the first, third and sixth months of mothers who were followed up with multidimensional visits after birth were significantly higher in the intervention group than in the control group. At one study emphasized that it is useful to emphasize the physical and psychological benefits of breastfeeding, as well as the health and bonding benefits, as a way to encourage more women to initiate and continue breastfeeding, and that it will be especially effective in groups that care more about body image, such as young mothers, where breastfeeding rates are low. At one study that breastfeeding mothers spend less time sleeping than non-breastfeeding mothers and that for optimal breastfeeding, the mothers paid or unpaid workload should be shared with other household members in the months after birth, thus meeting the mothers sleep needs. In a systematic review examining the effectiveness of perinatal breastfeeding support that included fathers/partners, it was determined that the inclusion of fathers in the process was associated with improved breastfeeding initiation rates and breastfeeding duration. Another systematic review suggested that there was a negative relationship between maternal anxiety in the postpartum period and the initiation and duration of breastfeeding. One study reported that exclusive breastfeeding rates increased significantly with privacy. In the presented studies, it was determined that various interventions were made and recommendations were made to increase breastfeeding rates. However, it was seen that there was a need for studies in which the needs of mothers regarding breastfeeding problems were addressed holistically and support was provided in line with their needs. It is obvious that in order to increase breastfeeding success and ensure the continuity of effective breastfeeding, a holistic assessment of mothers breastfeeding problems, determination of physical, psychospiritual, sociocultural and environmental factors that may cause deterioration in comfort and provision of comfort-focused nursing support are required.

Comfort in nursing practices consists of the process of defining the comfort needs of the patient, family or society, taking measures for their needs, evaluating the basic comfort level and the comfort level after the application. Kolcaba stated that comfort is a positive, holistic, multidimensional, theoretically definable and applicable concept as a result of his studies on the use of the concept of comfort in the nursing discipline. The Comfort Theory, developed by Kolcaba, is a nursing model that enables person-specific problems to be seen more systematically and to make plans for problem solving more easily. The aim of the model is to meet the physical, psychospiritual, sociocultural and environmental health care needs of the individual and to improve the comfort level and health outcomes. The taxonomic structure of the comfort theory is addressed in two stages. In the first stage, comfort levels are defined as relief, relaxation and superiority, taking into account the status of meeting individual comfort needs. Kolcaba states that when peoples needs are met, the feeling that emerges in people is relief; After the individuals needs are met, the individual will experience calmness, peace and contentment, resulting in a state of relaxation, individuals whose comfort needs are fully met will be able to overcome their problems (superiority). In the second stage, based on a holistic perspective, the dimensions of comfort are defined as physical, psychospiritual, sociocultural, and environmental. Physical comfort, includes physiological factors such as nutrition, excretion, elimination, rest, sleep, oxygenation status and pain that affect the individuals physiological state. Psychospiritual comfort, constitutes the individuals cognitive, emotional and spiritual components, and includes feelings related to being valued, self-concept and self-awareness. Environmental comfort, includes concepts related to the patients external environment, such as order, silence, comfortable objects, minimum odor, appropriate temperature, appropriate light and the view from the window. Sociocultural comfort, includes practices such as benefiting from economic support systems and providing information and consultancy.

In the literature review, positive effects of nursing care based on Kolcaba's Comfort Theory on care outcomes were demonstrated for adult cardiac patients, hospitalized elderly individuals, veterans, multiple sclerosis patients, adults with acute chest syndrome due to sickle cell disease, hemodialysis patients, patients in the preoperative period, breast cancer patients in palliative care, patients with cervical cancer, women undergoing hysterosalpingography, mothers who are about to give birth, mothers who have just given birth, and mothers who have had cesarean sections. In addition, it was seen that the scales named The Care in Obstetrics: Measure For testing Satisfaction COMFORTS Scale, General Comfort Scale, General Comfort Scale Short Form, Hemodialysis Comfort Scale, Nurse Comfort Questionnaire, Comfort Scale in Psychiatric Patients, Prenatal Comfort Scale, Birth Comfort Scale and Postpartum Comfort Scale were developed based on Comfort Theory. When the studies in which the Comfort Theory was used in the field of pediatric nursing were examined, it was determined that the theory was planned for; children with cerebral palsy and their parents, circumcised children and their parents, pediatric oncology patients and their mothers, newborns with Harlequin Ichthyosis, babies in the last period of their lives, children in intensive care, children in the postoperative period, children who underwent procedural procedures, interventions during labor, the mother's comfort and the effects on the newborn. However, the Comfort Theory was not applied to breastfeeding mothers. There is no study based on this. Kolcaba, theorist, was contacted via e-mail to get his opinion on this subject and Kolcaba gave a supportive feedback saying: I think your breastfeeding topic fits perfectly with the Comfort Theory. In addition, it was seen that there are scales called The COMFORT Behavior Scale, Premature Baby Comfort Scale, Newborn Comfort Behavior Scale and Kangaroo Care Comfort Scale in the field of pediatric nursing, but no measurement tool was found for the comfort of breastfeeding mothers.

When the literature is examined, it is seen that various current methods are used in breastfeeding support. In three different systematic reviews, web-based breastfeeding support, one of these methods, is emphasized as effective and useful in increasing breastfeeding self-sufficiency and sustainability. Reported in n a quasi-experimental study that mothers who received Web-based breastfeeding education had higher mean breastfeeding knowledge scores and more positive attitudes towards breastfeeding than those who did not. In two different randomized controlled studies, it was noted that Web sites were frequently used by mothers and their partners for breastfeeding support and that a Web-based breastfeeding education program could contribute to the development of breastfeeding self-efficacy. When the studies conducted in our country are examined, it has been observed that breastfeeding support is provided to mothers through the WhatsApp messaging application, online education and peer support, online education and telehealth application. However, no study has been found in which web-based interactive breastfeeding support is provided.

Despite many proven benefits for mothers and babies, breastfeeding rates are below the targeted rates in the world and in our country. It is clear that in order to increase breastfeeding rates, new approaches are needed to evaluate mothers holistically, to meet their individual needs that prevent breastfeeding based on scientific foundations and to support breastfeeding in this direction. In this project, determining the physical, psychospiritual, sociocultural and environmental comfort needs of mothers based on Kolcabas comfort theory to increase maternal comfort during breastfeeding, providing holistic breastfeeding support to mothers in line with their individual needs and including spouses/relatives in the support program can provide significant benefits in terms of child, mother and therefore public health.

In this context, the aim of the study is to determine the effect of breastfeeding support structured according to Kolcabas comfort theory given to mothers in the postpartum period on mothers breastfeeding comfort, and also the second aim is to develop the Postpartum Breastfeeding Comfort Scale and test its validity and reliability.

ELIGIBILITY:
Inclusion Criteria: • Primiparous mothers who are over 18 years of age and have given birth vaginally,

* Having a nuclear family structure,
* Living in the same house with their spouse,
* Having a medium socioeconomic level,
* The mother and baby are healthy,
* Not having sensory losses such as vision or hearing,
* Not having a diagnosed psychiatric history,
* Being able to read and write Turkish,
* Being open to communication and cooperation,
* Being a volunteer to participate in the research.

Exclusion Criteria: •Bebeğin kaybı,

* Annelerin postpartum süreçte travmatik bir durum yaşaması (bu durumdaki annelerle çalışma devam edecek ancak anneler analize alınmayacak),
* Kolcaba'nın Konfor Kuramına göre yapılandırılmış emzirme desteğine %70 katılmamış olmak

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breastfeeding mothers
Enrollment: 68 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of breastfeeding comfort in the study and control groups | Pre-test on postpartum day 0
  The Postpartum Breastfeeding Comfort Scale, which will be developed within the scope of the study, has a total of 49 items in the scale focusing on mothers' breastfeeding comfort. The scale is a 5-point Likert type and each item is scored between 1 and 5. A high score obtained from the scale indicates a high breastfeeding comfort level.
Evaluation of breastfeeding comfort in the study and control groups | Post-test at 6-8 weeks postpartum
  The Postpartum Breastfeeding Comfort Scale, which will be developed within the scope of the study, has a total of 49 items in the scale focusing on mothers' breastfeeding comfort. The scale is a 5-point Likert type and each item is scored between 1 and 5. A high score obtained from the scale indicates a high breastfeeding comfort level.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
can be published after the work is completed.